CLINICAL TRIAL: NCT02142491
Title: Pilot Project on Clinical Tolerance to a Live Attenuated Vaccine Against Influenza (Flumist®) in the Context of Influenza Vaccination in a Population Allergic to Eggs.
Brief Title: Clinical Tolerance to a Live Attenuated Vaccine Against Influenza (Flumist®) in a Population Allergic to Eggs
Status: Completed | Type: Observational
Sponsor: St. Justine's Hospital (Other)
Collaborators: Institut National en Santé Publique du Québec (Other)
Responsible Party: Principal Investigator, Dr. Anne Des Roches, M.D., Allergist, St. Justine's Hospital
Other Study IDs: FluMist240713
Record Dates: First submitted 2013-10-25; First posted 2014-05-20 (Estimated); Last update posted 2014-05-20 (Estimated); Status verified 2014-05

CONDITIONS: Egg Allergy
Keywords: Egg allergy; live attenuated influenza vaccine
MeSH Terms: conditions — Egg Hypersensitivity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The objective of this study is to verify the clinical tolerance to the vaccine Flumist (intranasal live attenuated influenza vaccine) in a population of egg allergic children. More specifically, the investigators want to estimate the risk of severe allergic reaction arising within 24 hours following the vaccination of egg allergic with Flumist.

DETAILED DESCRIPTION:
TITLE: Clinical tolerance of a live, attenuated influenza vaccine (FluMist®) in the context of influenza immunization in a population of egg-allergic children: A pilot project. Protocol #: FluMist240713.

1. INTRODUCTION

   In Canada, the flu vaccine is indicated for all children between 6 and 23 months of age. Epidemiologic and clinical studies have demonstrated that these children have a higher risk of complication and a higher rate of hospitalisation due to influenza. Trivalent inactivated influenza vaccines (TIV), which are administered intramuscularly, have long been used for preventative vaccination in this population. FluMist® is a live attenuated influenza vaccine (LAIV) administrated intranasally, which has been approved for use in Canada since 2010[1 ]. Besides avoiding the inconvenience and the anxiety related to intramuscular vaccines, FluMist® offers a better protection against influenza than the TIV. The Canadian National Advisory Committee on Immunization (NACI) recommends the preferential use of LAIV over TIV for influenza immunization in children 24 months old and over. Furthermore, LAIV use is favoured for children with chronic disease and those suffering from non-severe asthma [ 2].

   The influenza vaccine is manufactured using chicken egg embryos and as such, contains minimal residual quantities of ovalbumin (egg protein). In patients with an egg allergy, numerous clinical studies have demonstrated that its administration is safe with very little risk of anaphylactic reaction. Therefore, egg allergy is no longer a contra-indication to receiving TIV and these patients can now receive this vaccine without further precautions in CLSCs and doctors' offices[3 ,4 ]. There are no studies on the safety of LAIV administration in egg-allergic patients. As egg-allergic patients often have other atopic related comorbidities such as asthma, the increased protection against influenza which can be achieved with LAIV is desirable. The egg protein content in LAIV is comparable to that in TIV and its administration is intranasal rather than systemic. Therefore, it is reasonable to hypothesize that LAIV administration in egg-allergic patients is as safe as TIV administration in this same population. Yet, before recommending LAIV in egg-allergic patients, a study on its safety in this population is essential.

   1.1 Use of eggs in the production of influenza vaccines

   Because viruses are obligate intracellular parasites, vaccines against viruses must be produced using human or animal cells. Influenza vaccines currently used in Canada are produced by allowing the virus to multiply in chicken egg embryos. Despite rigorous purification processes, these vaccines, including Flumist®, still contain low residual quantities of ovalbumin (egg protein). The quantity of residual ovalbumin differs, at times significantly, between the different commercial influenza vaccines available in Canada, but also between different lots of the same vaccine [3]. While manufacturers have to assure that the influenza vaccines destined for the Canadian market do not contain more than 0.24 µg/dose of residual ovalbumin[ ], they are not required to divulge the final quantity. For this reason, a theoretical risk of anaphylaxis or hypersensitivity still exists in egg-allergic patients. However, the real risk of an anaphylactic reaction after an intramuscular influenza vaccination in an egg-allergic patent is quite low[1].

   1.2 Prevalence and clinical presentation of egg allergy

   Egg allergy is one of the most common food allergies[6]. Studies have demonstrated that 1 to 2% of young children could be allergic to eggs, which represents approximately 800 children in the 12 to 23 month age group in Quebec[7 ,8]. This allergy is often diagnosed around 18 months of age, when egg is introduced into the child's diet. Almost half of egg-allergic children are identified around 10 months of age[9 ,10 ]. We estimate that this allergy will have completely disappeared by the age of 5 in 66% of allergic children and 7 years of age in by 75%[11 ,12 ]. In the last decades, the duration of egg hypersensitivity seems to have increased until late childhood and sometimes into adolescence[13 ]. Persistent egg allergy into adulthood is rare. Persistent egg allergy essentially remains a paediatric issue. We can, therefore, estimate that in Quebec, there are over 3000 egg-allergic children between 1 and 9 years of age.

   The clinical presentation of egg allergy varies significantly. The signs and symptoms of IgE mediated allergic reactions can touch many systems and can have variable intensity, ranging from mild to severe. Symptoms can occur within a few minutes to several hours after ingestion of an egg-containing product, but the majority of allergic reactions occur within 30 minutes of contact[9]. The incidence of severe allergic reactions (anaphylaxis) to eggs is rare. We estimate that 7 to 10% of all declared anaphylactic reactions are due to egg protein[14 ].
2. SAFETY OF VACCINES IN EGG-ALLERGIC PATIENTS

2.1 Safety of the influenza vaccine in egg-allergic patients

In 1976, an outbreak of porcine H1N1 influenza A was observed in American army recruitment camps in Fort Dix, New Jersey. Despite this outbreak being relatively limited to recruitment camps, American health authorities implemented, in the general population, a massive vaccination campaign against this influenza strain. Before being abruptly stopped because of an increase in the number of cases of Guillain-Barre syndrome, over 48 million people had been vaccinations against this disease. Jointly to the mass vaccination campaign, the CDC had implemented a national surveillance program for post-vaccination side effects and had only 11 cases of post vaccination anaphylaxis registered. None of these cases occurred in egg-allergic patients. However, we are unaware of the number of people vaccinated who had an egg allergy, which limits the scope of the observed results.

Studies completed thereafter in egg-allergic children tended to demonstrate that this vaccine could safely be administered. A review of the literature of 27 studies prior to 2012 (table 1) consisting of 4172 egg-allergic patients vaccinated with TVI was published by our group[3]. Amongst these patients, no cases of severe allergic reactions were observed. The most common observed allergic reactions were mild (local erythema, local or distal urticaria, mildly wheezy breathing), though 1 patient did present generalized urticaria.

Since then, some other studies on this subject have been published. More specifically, the study by Greemhawt et al[15 ] demonstrated via retrospective and prospective cohorts, the safety of single dose TIV vaccination in severely egg-allergic patients.

Finally, a multicenter study conducted by our group over 5 influenza vaccine seasons permitted a better estimate of the risk of allergic reaction. Four hundred and fifty-seven doses of trivalent inactivated influenza vaccine were administered to 367 patients of which 132 (153 doses) reported a severe allergic reaction to eggs[4]. Four patient reported possible mild reactions secondary to previous influenza vaccines (1 urticaria, 2 vomiting and 1 eczema), but no severe allergic reactions were observed during the study. Thirteen patients developed mild allergic appearing symptoms in the 24 hours following vaccine administration but none of the 367 patients developed an anaphylactic reaction. Using a 95% confidence interval (Clopper-Pearson exact CI), the obtained results of this study allowed us to estimate a risk of anaphylaxis between 0 and 0.08% (0 to 1 on 1250 doses) for global population of egg-allergic patients and between 0 to 0.62% (0 to 1 on 161 doses) for patients with history of severe allergic reaction to eggs.

Following this study, the Quebec immunisation protocol (PIQ) was amended and now permits the administration of the influenza vaccine in egg-allergic patients in a single dose and in usual vaccination centers. Since these changes were implemented in the PIQ, no cases of anaphylaxis or death have been reported in this population.

2.2 Safety of LAIV (Flumist®)

Two formulations of FluMist® have been studied worldwide: a frozen (0.5ml/dose) and a refrigerated (0.2ml/dose). These 2 formulations are produced from the same viral strains and have a comparable degree of clinical efficacy. However, only the refrigerated (0.2ml/dose) formulation is authorised for use in Canada.

FluMist® is composed of attenuated viruses which cannot replicate at the temperature of the nasal mucosa. The most often reported side effects are nasal congestion and rhinorrhea.

Since people receiving this vaccine can excrete the virus in their nasal secretions in the days following vaccination, it is recommended to avoid this vaccine in immunocompromised patients and healthcare workers who are in contact with immunocompromised patients. Furthermore, it is recommended to avoid this vaccine in patients with severe asthma (defined as an individual on oral corticosteroid therapy or on high dose inhaled corticosteroids or an individual with wheezing on auscultation) (see section 3.4) and egg-allergic patients (see section 3.3).

2.3 Safety of LAIV (Flumist®) in egg-allergic patients: risk associated with a potential allergen administered intranasally

When the quantity of residual ovalbumine was measured by independent laboratories, only very low quantities were found, ranging between 0.00013 to 0.0017 µg per 0.2ml dose. The quantity of egg protein found in the intranasal vaccine is therefore, similar to that found in the TVI.

Given the different mode of administration between the TIV and the LAIV (intramuscular versus intranasal), it is important to underline the potentially different absorption of ovalbumin and its impact on the risk of an allergic reaction. Some studies have analyzed the absorption and the physiologic response when a food allergen is administered intranasally. More specifically, Clark et al[16 ] used the method of intranasal peanut provocation in allergic patients to evaluate the thermographic changes in nasal temperature. In their double-blinded provocation study, 10 µg of sterilized peanut extract was used for a nasal provocation and among the 16 patients, none presented systemic symptoms. Taking into account that the quantity of ovalbumin in LAIV is usually less than 0.24 µg per dose[1], and that the theoretic dose of food allergen is 40 times higher in the Clark et al study, the risk of an allergic reaction associated with the administration of LAIV in a egg-allergic population seems very low.

Moreover, when the systemic absorption of intranasally administered medications is compared to their oral form, it is much less important[17 ]. Ratner et al[18 ] demonstrated that the absorption of beclomethasone was approximately four times less than when administered intranasally. The quantity of ovalbumine which will truly be absorbed is probably significantly less than 0.24 µg contained in the LAIV.

2.4 Safety of Flumist® in asthmatic patients

Unlike American recommendations which suggest to avoid LAIV in all asthmatic patients[19 ], the National Advisory Committee on Immunization (NACI) of the Public Health Agency of Canada (PHAC) recommends this vaccine in asthmatic patients except those with severe asthma defined as asthmatic individuals on oral corticosteroids or on high dose inhaled corticosteroids or asthmatic individuals with wheezing on auscultation[4].

Unlike American recommendations, Health Canada recommendations are based on more recent studies. Many studies have demonstrated the efficacy and the safety of using LAIV in a population of moderately to severely but stable asthmatic individuals. In 2003, Flemming et al[20 ] demonstrated in 2000 asthmatic children and adolescents a better efficacy of LAIV as well as an asthma exacerbation rate similar to TIV. Furthermore, Redding et al[21 ] studied the safety of LAVI in 1997 with 48 patients between 9 to 17 years old with moderate to severe but stable asthma. The percentage of change in forced expiratory volume (FEV1) evaluated up until the fifth day was similar between the vaccinated and the placebo group (0.2% versus 0.4%, p=0.78).

2.5 Intradermic testing with the flu vaccine

Intradermic testing with the flu vaccine does not detect egg-allergic patients who are at greater risk of developing an allergic reaction after administration of the flu vaccine. Therefore, its use in not recommended[22 ].

3. AIM

The aim of this study is verify the clinical tolerance of the inactivated, attenuated flu vaccine (Flumist®) in an egg-allergic population. More specifically, we will estimate the risk of severe allergic reactions in the 24 hours following vaccination with Flumist® in egg-allergic patients.

4. METHODS

4.1 Population :

4.1.1 Case group

4.1.1.1 Inclusion criteria

Children between 2 and 17 years of age with a confirmed egg allergy and for whom the flu vaccine is indicated because they are considered at high risk or because they desire protection against the flu virus.

4.1.1.2 Confirmation of an egg allergy

Confirmation of an egg allergy requires a set of criteria which vary depending on whether or not they have ever eaten eggs.

4.1.1.3 Patients having already eaten eggs must meet the following 2 conditions:

1. Patients must have experienced in the 60 minutes following ingestion one of the signs or symptoms listed below:

   Mild sings/symptoms:

   1) Cutaneous pruritis or mild urticaria (less than 5 urticarial plaques) or erythema 2) Rhinorrhea, sneezing or nasal congestion 3) Pruritis, erythema, edema or tearing 4) Throat or palate pruritis 5) Dyspnea (not objectified) 6) Vomiting or diarrhea

   Moderate to severe signs/symptoms:
   1. Facial angioedema
   2. Systemic urticaria (more than 5 urticarial plaques)
   3. Objectified dyspnea or respiratory distress
   4. Wheezy breathing
   5. Cough
   6. Weakness or altered level of consciousness
   7. All other reactions requiring administration of epinephrine
2. confirmation of the allergy by one of the following methods within 6 months of the reaction:

   1. a positive egg skin prick test (diameter of induration > 3 mm more than the negative control (saline) read 10 to 15 minutes after the procedure).
   2. a specific egg IgE level >0.35 kIU/L

4.1.1.4 In patients never having consumed eggs or egg containing products or with an uncertain clinical history of reaction to eggs, the diagnosis must be confirmed by the following 2 methods in the 6 months following the reaction:

1. a positive egg skin pric test and
2. a specific egg IgE level measured by ImmunoCAP of: > 2kIU/L in children less than 2 years old or > 7kIU/L in children 2 years old and over.

4.1.1.5 Exclusion criteria

We could not vaccinate patients with the following conditions. However, some of these conditions can be temporary as they are reversible. Therefore, vaccination must be done at a moment when the situation has improved.

Exclusion criteria:

1. poorly controlled asthma on the day of vaccination defined by the presence of wheezy breathing and/or cough at the time of vaccination or wheezing on auscultation;
2. severe asthma defined as an individual on oral corticosteroids or on high dose inhaled corticosteroids;
3. the presence of an urticarial rash on physical exam;
4. the use of antihistamines (first or second generation) 3 to 7 days (respectively) before vaccination;
5. the presence of a moderate to severe acute illness (with for example, fever, irritability, inconsolable crying, lethargy, abnormal fatigue, vomiting, diarrhea, pallor, cyanosis or diaphoresis);
6. immunocompromised patients and healthcare workers in contact with immunocompromised patients.

4.1.2 Control group

100 individuals without a history of egg allergy, never having received the intranasal flu vaccine will be recruited. These control subjects will be recruited in a manner to allow a similar age distribution to the allergic patients.

4.1.2.1 Inclusion criteria

Children between 2 and 17 years of age without a history of egg allergy and for whom there is an indication for the flu vaccine because they are considered at risk for complications or because they desire a protection against the flu virus.

4.1.2.2 Exclusion criteria

They are the same as in the case group. See section 4.1.1.5.

4.1.3 Identification of patients

Allergic patients will be contacted starting in October to inform them of this project. This will include:

1. Known allergic patients who will be contacted by their allergists themselves;
2. Patients of pediatricians and general practitioners who have been informed of the project and who will have been referred;
3. The department of allergy and immunology will sent to known egg-allergic patients a letter informing them of the project and inviting them to take an appointment at the clinic. These patients will be identified by, among other things, lists of positive egg specific IgE levels done in the last 24 months;
4. As needed, an ad for the project, in written media or electronically, could be used.

Controls will be recruited at the allergy clinic at Ste-Justine hospital. These patients may be followed for allergies but will not have an egg allergy. Controls may also be recruited by ads in social media or by other services.

4.2 Clinical procedures

On the vaccination day, participants will have to follow the procedure below:

1. A research nurse will explain to the parents of the participants what is to be expected in the context of this project. She will ask the patients to read the consent form for the project. She will mention that there will be a follow-up by telephone 24 hours after the vaccination to ask about the clinical status of the child. Those who accept will have to sign the consent form. If they do not accept, they will be vaccinated using TIV according to the current recommendation of Quebec public health.
2. In the context of the clinical approach of our service, parents will fill out an auto-administered questionnaire on the clinical history of their child's egg allergy. This questionnaire will take approximately 15 minutes to complete. The allergist will verify the answers with the parents and will proceed to examine the child including an examination of the skin and pulmonary auscultation at most 30 minutes prior to vaccination. For the control subjects, the physical exam will also be done by the allergist in the clinic.
3. For children with an egg allergy, a clinical revaluation (skin prick test and egg specific IgE levels by ImmunoCap) will be done if the latest values are more than 6 months old or if they are not adequately documented. This test will take approximately 15 minutes.
4. The vaccine used will be the live, attenuated influenza vaccine (LAIV) i.e Flumist® by AstraZeneca. As the egg allergen (ovalbumin) content in LAIV is comparable to the intramuscularly administered vaccine and that the risk of allergic reaction with TIV has been shown to be very low when administered in a single dose, the intranasal vaccine Flumist® will be administered by the nurse or doctor in a single dose of 0.2ml intranasally, as recommended by the manufacturer. This vaccination will be followed by a 60 minute observation period. We will examine the child 60 minutes after vaccination and at any time if the child, parent or personnel suspects an allergic reaction or adverse effect.

   The wait time after the vaccination will occur in the waiting room of the allergy clinic under the supervision of a nurse. We will ask the parents and the child to inform the doctor or the nurse if they observe any of the following manifestations: erythema, pruritis, rash, sneezing, rhinorrhea, tearing, nasal congestion, voice change, cough, difficulty breathing, noisy breathing, pallor, weakness, vomiting or diarrhea. We will ask them to also advise the members of the research team of any other reactions or concerning states.
5. Before leaving, parents will be questioned on the presence of allergic symptoms.

   If a reaction occurs, it will be treated based on the allergist or supervision doctor decision. The allergy clinic where vaccination will occur is equipped with the necessary material to treat an allergic reaction i.e. epinephrine, oral and injectable diphenhydramine, inhaled salbutamol, oral and intravenous corticosteroids and oxygen.
6. Telephone follow-up

   All parents will receive an emergency phone number to contact in case of allergic reaction within the 24 hours following vaccination. This will be the contact information of the principal investigator of the project, Dr Anne Des Roches, or the allergist on call if she is absent. Moreover, the phone number will also be provided to the telephonists of Ste-Justine Hospital who can call Dr Des Roches or the allergist on call. She (or he) will evaluate the patient for a biphasic reaction or for a delayed reaction or could have the patient come to the allergy clinic or refer the patient to the emergency department according to the situation. Parents will be advised to contact emergency services first if there is a severe delayed reaction.

   Parents will be called the following day to enquire about the presence of any allergic manifestation that could have appeared in the 24 hours following vaccination.

   4.2.1 Second dose

   Children between 2 and 8 years of age, who have never received a trivalent seasonal flu vaccine and who have tolerated the first dose, will be invited to a second appointment to receive a booster dose, 1 month later. The second dose will be followed by on observation period of 15 minutes.

   4.3 Sample size

   As this is a pilot project, we aim to recruit of 100 egg-allergic patients and 100 control patients. According to the results, a multicentre study on a large number of egg-allergic patients could be done at a later time.

   4.4 Primary outcome and statistical analysis

   The primary outcome will be the presence of anaphylactic reactions following flu vaccination with LAIV. An anaphylactic reaction will be defined according to the Brighton Collaboration criteria, an international organization that standardises the criteria defining vaccine side effects[23].

   Secondary outcomes will be the presence of all allergic manifestations as described in section 4.1.1.3 within the 24 hours following flu vaccination.

   We will compare the proportion of patients and control presenting allergic symptoms using the exact Fisher test. We will estimate the risk of anaphylaxis and its 95% confidence interval using the Clopper-Pearson exact method.

   4.5 Schedule and surveillance of the study

   This study will be conducted over a period of 6 months, i.e. from October 2013 to March 2014, which corresponds to the flu vaccination period.

   An analysis of the data pertaining to anaphylactic reaction will be compiled regularly by the study's principal investigator.

   The study will cease if one of the following situations occurs during the study:
   * if a child develops fatal or almost fatal reaction;
   * if more than 2% of children develop reactions requiring epinephrine administration.

     5. Risks and benefits of the study

   For egg-allergic patients who desire the flu vaccine, the risk of participation in this study is the risk of developing an allergic reaction following Flumist® vaccination.

   Although nasal congestion, rhinorrhea and cough are the most common reported side effects in patients receiving this vaccine, if an allergic reaction occurs, it could manifest as more important nasal symptoms (congestion, rhinorrhea, pruritis, sneezing, edema), as well as oral symptoms or systemic symptoms, accompanied by pruritis, urticaria, wheezy breathing or, in severe cases, hypotension, throat swelling or tightness and/or difficulty breathing. An allergic reaction can also present as nausea, abdominal pain and/or sudden vomiting. Patients will be monitored closely during the whole procedure, as well as in the hour following it for the onset of these symptoms. If need be, they will be seen by the study doctor who will evaluate the need for antihistamines, epinephrine, corticosteroids or who will institute specialized techniques to maintain vital functions. The risk of a severe reaction is probably very low considering the low egg content in the vaccine.

   For the control group, there is no additional medical risk to participating in this study, as they will be receiving the seasonal flu vaccine in the same manner that they would if they were not participating in the study and no supplemental procedure will be necessary except for an observation period of 60 minutes, a follow-up telephone call 24 hours after vaccination and a short medical questionnaire.

   Aside from a more stringent observation for reactions to the vaccine, controls will not encounter any direct benefits to their participation in this study. For the case participants, the intranasal flu vaccine will allow them to obtain a better protection against the seasonal flu vaccine than received with TIV.

   Furthermore, if the results obtained confirm the safety of FluMist® in egg-allergic patients, this will allow reassurance of healthcare professional of the safety of vaccination in egg-allergic patients. More long term, this will allow egg-allergic patients to receive the LAIV rather than being limited to TIV.

   6. Medications under investigation The FluMist® vaccine made by AstraZeneca will be provided and routed to Ste-Justine Hospital by the National Institute of Public Health under the specific storage conditions set by the manufacturer. The vaccines will be under the conditions required by the manufacturer in the Ste-Justine research center, under the responsibility of the principal investigator. The Ste-Justine research center is equipped with a refrigerator with temperature control monitors, allowing for verification of all changes in temperature which can then be reported to the principal investigator. Vaccines will be stored in a safe and secure environment. Information pertaining to the arrival of the vaccines, the doses administered and the return or destruction (if warranted) of the vaccines will be documented.

   7. Protection of data

   The data compiled from this study will be anonymized and entered into an Excel database. The database will be kept on a Ste-Justine computer which can only be accessed by the research team. The computer is username and password protected and is situated in a locked office.

   8. Adverse reactions to medication report In this study, Canadian regulations will apply for the reporting of serious adverse effects. For medications used in the context of clinical trials in Canada, only serious and unexpected adverse effects must be rapidly reported to Health Canada.

   Serious but expected adverse effects and serious therapeutic incidents observed during the clinical trial but not considered secondary to the product in question, whether they are expected or not, do not require expedited reporting.

   A report will be completed in the following cases:

   - in the 15 days following the moment when the situation if known, if the effect is not fatal but puts the patient's life in danger;

   - as soon as possible in the 7 days following the moment when the situation if known, if death occurs or if the effect can put the patient's life in danger;
   * in the 8 days following the notification of Health Canada of adverse effects, a detailed report containing an estimation of the importance of the repercussions and findings.

   Each case of adverse effects subject to expedited declaration will undergo a distinct declaration consisting of the all the elements required in Health Canada guidelines/ICH E2A: Clinical Safety Data Management: Definitions and Standards for Expedited Reporting.

   Data pertaining to the harmlessness of a medication will be communicated in an ongoing process to the research ethics committee.

   9. Surveillance of data security committee

   A committee to monitor the security of the collected data shall be formed by professionals who are not implicated in the elaboration of this protocol. The regulations set out by Health Canada shall be followed.

   The primary responsibilities of this committee shall be the following:
   1. Periodic meetings (approximately every 2 months or more if necessary) to evaluate the study results in respect to security, the management of the study and the progress of recruitment.
   2. To elaborate recommendations on the continuation, modification or cessation of the study.
   3. To evaluation compiled serious adverse effects.

   10. Ethics Parents who do not wish to sign the consent form can get their children vaccinated with TIV according to the regular clinical protocol as recommended by Quebec public health.

   The information and consent forms will explain to the control group that they must remain in the clinic for a longer period of time after vaccination then would be normally required (60 versus 15 minutes) and that they will have to fill out a short medical questionnaire as well as receive a follow-up phone call.

   The safety of patients will be assured by providing vaccination in a center equipped with all the necessary material and personnel to rapidly respond to an anaphylactic reaction, rapid access to an emergency department and close observation.

   Questionnaire will only identified by number and only this number will be used in the database to ensure confidentiality.

   11. Schedule

   June 2013 Submission to the ethics committee

   30 October 2013 Start of vaccination

   12. References: Available upon request

ELIGIBILITY:
Inclusion Criteria:

* Egg allergic children

Exclusion Criteria:

* Uncontrolled asthma the day of immunization
* severe asthma treated by oral steroids or high dose of inhaled steroids
* urticaria on the day of immunization
* antihistamines taken in the previous 3 to 7 days of immunization
* acute disease on the day of immunization (fever,irritability, vomiting, diarrhea, pallor, cyanosis, diaphoresis, lethargy)
* immunosuppressed patients or health worker who should be in contact with immunosuppressed patients.

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The population will be a group of 75 egg allergic children (2 to 17 years old) and a group of 75 non-allergic children (2 to 17 years old). Egg allergic children will be selected from the allergy clinic of a university children hospital and non-egg allergic children will be selected from the community.
Sampling Method: Non-Probability Sample
Enrollment: 124 (Actual)
Dates: Start 2013-11; Primary Completion 2014-02 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Anaphylactic reaction following the administration of the vaccine | Observation period at hospital during one hour post vaccination. And Follow-up phone call 24 hours post vacciation.

SECONDARY OUTCOMES:
Allergic reactions occuring in the 24 hours following the immunization with Flumist. | Datas will be assessed following the period of immunization. 24 hours following the immunization

CONTACTS AND LOCATIONS:
Overall Officials: Anne Des Roches, MD, Principal Investigator — St. Justine's Hospital; Gaston De Serres, MD, Principal Investigator — Santé Publique du Québec
Locations (1):
- CHU Sainte-Justine, Montreal, Quebec, Canada